CLINICAL TRIAL: NCT02377726
Title: Internet Based Treatment for Alcohol Dependence Among Anonymous Help Seekers on the Internet : A Randomized Controlled Trial
Brief Title: Anonymous Treatment on the Internet for Alcohol Dependence: A Randomised, Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Public Health Agency of Sweden (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/1758-31-2
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Harmful Alcohol Use; Alcohol Use Disorder
Keywords: Randomized Controlled Trial; Alcohol; Internet; Internet based therapy; Cognitive behavioral therapy
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet self-help with support (Experimental): eChange Alkoholhjälpen is an internet based self help program consisting of 5 modules. Patients will have access to Alkoholhjälpen counselor support through secure comments at every module they complete.
  Interventions: Behavioral: Alkoholhjälpen counselor support; Behavioral: eChange Alkoholhjälpen
- Internet self-help (Experimental): eChange Alkoholhjälpen is an internet based self help program consisting of 5 modules.
  Interventions: Behavioral: eChange Alkoholhjälpen
- Information (Active Comparator): Brief information on resources that can be accessed through the open access website Alkoholhjälpen: Information on alcohol and health, where and how to find treatment and an internet discussion forum.
  Interventions: Behavioral: Alkoholhjälpen

INTERVENTIONS:
Behavioral: Alkoholhjälpen counselor support — Users will have access to counselor support through secure comments at the end of every module they complete in the self help program.
  Arms: Internet self-help with support
Behavioral: eChange Alkoholhjälpen — An internet based intervention program (iCBT) consisting of 5 modules. Fully automated self-help
  Arms: Internet self-help; Internet self-help with support
Behavioral: Alkoholhjälpen — A swedish, open access website that includes information on alcohol, on how to find treatment and an internet discussion forum
  Other Names: alcoholhjalpen.se, alcohol-help-site
  Arms: Information

SUMMARY:
Internet based self help program with or without support of a counselor is tested among anonymous Internet help seekers at an open access website.

DETAILED DESCRIPTION:
A 5 module Internet based self help program based on motivational interviewing and cognitive behavioral therapy is tested among anonymous Internet help seekers.The design is a three armed randomized controlled study, and outcomes are measured in terms of changes in alcohol consumption, problematic alcohol use, alcohol dependence alcohol use disorder, anxiety, as well as depression and quality of life. 2400 participants are recruited entirely online from an open access website. Consenting participants will be randomized into one of three groups: 1.Internet based self help program with counselor support, 2.Internet based self help program without counselor support or 3. Information about the open access websites resources: information on alcohol and health, where you can find treatment and a online discussion forum. Follow-up will be conducted online after 3, 6, 12 and 24 months in all three groups.

ELIGIBILITY:
Inclusion Criteria:

AUDIT-score >16 points and/or at least 3 criteria of alcohol dependence (ICD-10)

Exclusion Criteria:

Inadequate Swedish language skills No Internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) (Change in total in consumption of alcohol last 7 days) | 3, 6, 12 and 24 months
  Change in total in consumption of alcohol last 7 days

SECONDARY OUTCOMES:
Time Line Follow Back (TLFB) (Change in number of standard drinks per day during last 7 days) | 3, 6, 12 and 24 months
  Change in number of standard drinks per day during last 7 days
Time Line Follow Back (TLFB) (Change in number of consumption days during last 7 days) | 3, 6, 12 and 24 months
  Change in number of consumption days during last 7 days
Time Line Follow Back (TLFB) (Change in number of days binge-drinking days during last 7 days) | 3, 6, 12 and 24 months
  Change in number of days binge-drinking days during last 7 days
Alcohol dependence (ICD-10) (Change in number of criteria for alcohol dependence met) | 3, 6, 12 and 24 months
  Change in number of criteria for alcohol dependence met
Alcohol Use Disorder (DSM-5) (Change in number of criteria for alcohol use disorder met) | 3, 6, 12 and 24 months
  Change in number of criteria for alcohol use disorder met
Alcohol Use Identification Test (AUDIT) (Change in total AUDIT score, as a summarized measure of alcohol use) | 3, 6, 12 and 24 months
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems)
Montgomery Asberg Depression Rating Scale - Self report (MADRS-S) (Change in total MADRS-S score) | 3, 6, 12 and 24 months
  Change in total MADRS-S score, as a summarized measure of depression
Generalised Anxiety Disorder Assessment (GAD-7) | 3, 6, 12 and 24 months
  Change in total GAD-7 score, as a summarized measure of anxiety
The EuroQol generic health index (EQ5D) | 3, 6, 12 and 24 months
  Change in total EQ5D score, as a summarized measure of quality of life
Questions about help-seeking behavior | 3, 6, 12 and 24 months
  Change in help-seeking for alcohol related problems from professionals
Questions about help-seeking behavior (Change in help-seeking for alcohol related problems from family and friends) | 3, 6, 12 and 24 months
  Change in help-seeking for alcohol related problems from family and friends

OTHER OUTCOMES:
The Readiness Ruler (Scores between 0 and 100) | 3, 6, 12 and 24 months
  Scores between 0 and 100. In this study, "I am not ready to change my drinking habits" and "I am very much ready to change my drinking habits".
Use of Internet based program and website (Number of visits and number of completed exercises in the Internet based program and website) | From baseline to 3 months
  Number of visits and number of completed exercises in the Internet based program and website
Working alliance with internet based intervention (eSRS) (4 scale questions on the users alliance with the internet based intervention ) | 2 and 5 weeks
  4 scale questions on the users alliance with the internet based intervention (program and/or website)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Andreasson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Public Health Sciences, Stockholm, Sweden

REFERENCES:
- [Background] Sinadinovic K, Wennberg P, Johansson M, Berman AH. Targeting individuals with problematic alcohol use via Web-based cognitive-behavioral self-help modules, personalized screening feedback or assessment only: a randomized controlled trial. Eur Addict Res. 2014;20(6):305-18. doi: 10.1159/000362406. Epub 2014 Oct 4. PMID 25300885
- [Derived] Johansson M, Berman AH, Sinadinovic K, Lindner P, Hermansson U, Andreasson S. Effects of Internet-Based Cognitive Behavioral Therapy for Harmful Alcohol Use and Alcohol Dependence as Self-help or With Therapist Guidance: Three-Armed Randomized Trial. J Med Internet Res. 2021 Nov 24;23(11):e29666. doi: 10.2196/29666. PMID 34821563
- See also: Open access website — https://alkoholhjalpen.se
- See also: Berman's profile at Uppsala University — https://www.katalog.uu.se/profile/?id=N19-2760